CLINICAL TRIAL: NCT02617719
Title: Comprehensive Geriatric Assessment in Primary Care: The Fit for Late Life
Brief Title: Comprehensive Geriatric Assessment in Primary Care: The Fit for Late Life Project
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: b2xrypzt
Record Dates: First submitted 2015-11-18; First posted 2015-12-01 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Ageing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Primary care: Staff, patients aged 75 years and older and their carers associated with a single, participating United Kingdom primary care practice.

SUMMARY:
Comprehensive Geriatric Assessment is an effective process to identify and address the needs of older patients. In the United Kingdom this usually takes place in acute care or in the patients home. This project will assess the feasibility of implementing this service in primary care.

DETAILED DESCRIPTION:
With the ageing of the United Kingdom population, it is crucial that evidence on optimal healthcare is effectively translated into improved clinical practice to both maximise the health and independence of older people as well as contain costs. Comprehensive Geriatric Assessment (CGA) is a multidimensional, interdisciplinary process used to identify and address the complex healthcare needs of older people. Evidence of its effectiveness has been confirmed in a number of systematic reviews and meta-analyses and beneficial outcomes reported include improved function and independence. However its implementation across healthcare settings remains variable. This study aims to establish the feasibility, acceptability and cost of implementing a Comprehensive Geriatric Assessment Clinic in a single primary care practice.

The Fit for Later Life Project describes the implementation of a Comprehensive Geriatric Assessment Clinic in primary care for older people who referred by their General Practitioner (GP). We will utilise a mixed-methods design including Normalisation Process Theory (NPT), a sociological toolkit designed to explore how different stakeholders engage with the real-world process of translating evidence into practice. Interviews and focus groups will be used to collect data from patients, carers and health professionals on coherence, cognitive participation, collective action, and reflexive monitoring. These data will be thematically analysed to identify barriers, strengths and weaknesses for the implementation of a Comprehensive Geriatric Assessment Clinic in primary care. A clinical audit of the records of older people who are service users at the participating practice will be conducted and an assessment will be made of the costs of the clinic. Together these data will provide implementation guidelines describing the feasibility and acceptability of a United Kingdom primary care Comprehensive Geriatric Assessment clinic.

The planned outcome is guidelines for the implementation of a Comprehensive Geriatric Assessment Clinic in United Kingdom primary care. The barriers and facilitators that affect starting and running the service will be described as will the patients who could potentially attend and those who actually attend. The costs will also be determined.

This research is funded by the National Institute for Health Research Collaboration for Leadership in Applied Health Research and Care (NIHR CLAHRC) Wessex.

ELIGIBILITY:
Inclusion Criteria:

1. Involved in care of patient aged 75 years or older at the participating United Kingdom primary care practice.
2. Patient aged 75 years or older at the participating United Kingdom primary care practice.
3. Carer of patient aged 75 years or older at the participating United Kingdom primary care practice.

Exclusion Criteria:

1. Patient in end of life care
2. Patient does not have the mental capacity to act. -

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Staff: Primary care staff who are involved in the care of patients aged 75 years and older from a single United Kingdom primary care practice.
  Patients: Patients aged 75 years and older from a single United Kingdom primary care practice.
  Carers: Carers of patients aged 75 years and older from a single United Kingdom primary care practice.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Experience of the acceptability of a Comprehensive Geriatric Assessment clinic in United Kingdom primary care | 6 months
  Qualitative interviews performed before and after the new clinic where the participants describe their perceptions and experience of the the new Comprehensive Geriatric Assessment in United Kingdom primary care.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn N Lansbury, PhD, Principal Investigator — University of Southampton, UK

IPD SHARING:
Plan to Share IPD: Undecided